CLINICAL TRIAL: NCT01894542
Title: An 8 Week Study to Compare the Effects of Two Combinations of Water Soluble and Non-water Soluble Cod Residual Meals on Glucose Regulation in Overweight and Obese Adults
Brief Title: A Study of the Effects of Intake of Two Cod Residual Meals on Glucose Regulation in Overweight and Obese Adults
Acronym: FISK4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Granit AS Transport & Tourism (Other); Norwegian Seafood Center (Unknown); Nofima (Other)
Responsible Party: Principal Investigator, Oddrun Anita Gudbrandsen, PhD, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011/572-14
Record Dates: First submitted 2013-07-03; First posted 2013-07-10 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cod protein from presscake (Experimental)
  Interventions: Dietary Supplement: Cod protein from presscake
- Cod protein from presscake + stickwater (Experimental)
  Interventions: Dietary Supplement: Cod protein from presscake + stickwater
- Control (Placebo Comparator): Control group will receive tablet containing only tablet fillers (the same as in the cod protein tablets).
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Cod protein from presscake — 6g protein per day for 8wk
  Arms: Cod protein from presscake
Dietary Supplement: Cod protein from presscake + stickwater — 6 g protein per day for 8 wk
  Arms: Cod protein from presscake + stickwater
Dietary Supplement: Control
  Arms: Control

SUMMARY:
The investigators have previously shown the intact protein from cod filet improves glucose regulation and serum lipid profile in overweight adults. A large amount of trimmings from various fish species such as cod is thrown away or sold at very low prices for animal feed, and analyses of the amino acid composition reveals that this can be a good protein source for humans. Two fractions are normally isolated from intact fish meal, i.e. water soluble and non-water soluble proteins. In the present study the investigators will compare these fractions, by studying their effects on glucose regulation in overweight/obese adults.

DETAILED DESCRIPTION:
Participants receive 6g per day of water soluble on non-water soluble cod protein as tablets for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI>28
* healthy
* fasting blood glucose <7.0 mmol/L
* stable body weight with less than 5 kg fluctuation during the last 4 months

Exclusion Criteria:

* known disease or metabolic disturbances related to overweight or obesity
* use of prescription medications that affect blood glucose, blood lipids or inflammatory status
* allergies towards fish or seafood
* undertaking a weight loss diet
* tobacco use exceeding >15 cigarettes/day
* pregnancy or breastfeeding
* high seafood consumption
* use of dietary supplements including cod liver oil or other marine fatty acids
* allergies towards fish, milk, egg

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance | 8 weeks
  Serum glucose will be measured in fasting and postprandial state

SECONDARY OUTCOMES:
Gene expression | 8 weeks
  Changes in gene expression in adipose tissue related to the circulating markers of glucose regulation.
Amino acids and amino acid metabolites | 8 weeks
  Amino acids and amino acid metabolites will be measured in serum and urine
Comparisons of metabolites and co-factors involved in one-carbon metabolism in serum and urine | 8 weeks
  Concentrations of relevant metabolites and co-factors were measured in serum and urine

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bergen, Bergen, Norway

REFERENCES:
- [Background] Vikoren LA, Nygard OK, Lied E, Rostrup E, Gudbrandsen OA. A randomised study on the effects of fish protein supplement on glucose tolerance, lipids and body composition in overweight adults. Br J Nutr. 2013 Feb 28;109(4):648-57. doi: 10.1017/S0007114512001717. Epub 2012 May 31. PMID 22647247